CLINICAL TRIAL: NCT02953613
Title: LipiScan- Ultrasound INterrogation of Atherosclerotic Coronary Arteries: Correlations With Non-invasive Coronary Computer Tomographic Angiography. (LUNAR-CCTA Study)
Brief Title: LipiScan- Ultrasound INterrogation of Atherosclerotic Coronary Arteries:
Acronym: LUNAR-CCTA
Status: Terminated | Type: Observational
Why Stopped: unable to identify sufficient eligible patients to meet enrollment goals
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Ivan D. Hanson, MD., Corewell Health East
Other Study IDs: 2015-129
Record Dates: First submitted 2016-08-24; First posted 2016-11-03 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Cardiac Catheterization; Cardiac intervention; coronary angiogram; coronary artery disease; atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiac Catheterization with NIRS/IVUS: Cardiac cathetirization with NIRS/IVUS assessment if with blockage of indeterminate severity (greater or equal to 20% to 70%). One day to one week after invasive catheterization a CCTA will be done to correlate result, then CCTA will be repeated at 24 months
  Interventions: Device: NIRS/IVUS

INTERVENTIONS:
Device: NIRS/IVUS — Cardiac catheterization using infraredx
  Other Names: Infraredx

SUMMARY:
The goal of this study is to correlate both plaque and % lipid core content assessed by NIRS-IVUS (Imaging technique) to plaque burden and % lipid core content in coronary computerized tomographic angiography (CCTA) completed at 1 week in non-culprit coronary arteries.

DETAILED DESCRIPTION:
This is a prospective single center study that will enroll 200 patients undergoing clinically indicated cardiac catheterization for stable ischemic heart disease or unstable chest pain, who are also undergoing NIRS-IVUS direct coronary imaging of a culprit lesion based on routine clinical indications. The NIRS/IVUS catheter uses near-infrared light (red laser light) and intravascular ultrasound (sound waves) to identify fatty plaques in the coronary artery. Standard angiography, near-infrared spectroscopy (NIRS) and intravascular ultrasound (IVUS) are three widely used clinical methods to image narrowing within the coronary arteries at the time of cardiac catheterization.

Independently from this study, patients have agreed to a cardiac catheterization (angiogram - an x-ray picture of the heart) and possible angioplasty procedure and/or stenting as part of clinical care. During the cardiac catheterization if the blockage is bad enough an inflatable balloon attached to the end of a thin tube (called a catheter) is positioned in the narrowed part of the coronary artery. The balloon is then inflated, which opens the artery so that blood can flow more easily. After the balloon angioplasty procedure, a stent may be placed in the coronary artery. A stent is an expandable metal tube that helps to hold the artery open so that blood can continue to flow through the artery.

If the doctor determines that there are other blockages of indeterminate severity (≥20%-≤70% blockage) that require NIRS/IVUS assessment to better assess the severity of the blockage or that angioplasty and/or stenting is necessary the NIRS/IVUS catheter will be used. If severe non-culprit blockages are incidentally identified, they may be treated at the discretion of the operator. After the invasive coronary catheterization patients will follow Beaumonts standard post procedureal treatment guidlines.

Between one day and one week after the invasive catheterization patients will return for a research related non-invasive coronary Cat scan. A coronary Cat scan will be repeated at 24 months (2 years) to assess any of the blockages of indeterminate severity that were identified during your initial invasive cardiac catheterization. Upon arrival for Cat scan a nurse will ask the patient a few questions, insert a small tube in one of the patients arm veins. Blood will be drawn from the small tub and kidney function will be assessed. All Cat scans will be completed under Beaumont Hospital Institutional guidelines for coronary Cat scans. If significant blockages are identified, the patient may be notified to complete additional testing, which may include a stress test or a coronary angiogram. If other non-cardiac incidental findings are noted that require additional clinical or imaging follow up, the patient and the primary care physician will be notified.

A study doctor, nurse, or research coordinator will follow-up with each patient by phone six times over five years while participating in the registry. Phone calls will be performed at the following intervals from the date of the index procedure: 6 months (± 14 days); 12 months (± 30 days); 24 months (± 60 days); 36 months (± 60 days); 48 months (± 60 days); and 60 months (± 60 days) to ask patients how they are doing and to collect any major adverse cardiac events.

The Plan is for an enrollment period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable ischemic heart disease or ACS undergoing cardiac catheterization and possible PCI of a culprit lesion
* The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent approved by the Institutional Review Board.
* The study patient agrees to comply with all required post-procedure follow up.
* Patient age 18-89 years old

Exclusion Criteria:

* STEMI within the prior 24 hours
* Cardiogenic shock or hypotension needing inotropes or hemodynamic support device
* Intra-procedural complication (perforation or a complication that would necessitate immediate-unplanned revascularization) during index PCI procedure
* History of CABG
* Subject life expectancy less than 2 years at time of index catheterization
* Pregnant or unknown pregnancy status
* Psychological unsuitability or extreme claustrophobia
* Currently participating in another investigational cardiac device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials
* Inability to tolerate beta blockers
* Atrio-ventricular block (grade II-III), prolonged QT interval or sick sinus syndrome
* Renal insufficiency (creatinine ≥ 1.6 and/or, GFR < 60 ml/min) or renal failure requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to Beaumont Hospital for elective invasive coronary angioplasty and possible percutaneous intervention
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-04-28; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
To correlate blockages by NIRS-IVUS with CCTA | 5 years
  To correlate both plaque burden and % lipid core content assessed by NIRS-IVUS to plaque burden and % lipid core content on coronary computerized tomographic angiography (CCTA) completed at 1 week in non-culprit coronary arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Hanson, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No